CLINICAL TRIAL: NCT01128322
Title: A Randomized, Double-blind, Multi-center, Multi-factorial, Phase 2 Trial to Evaluate the Efficacy and Safety of S-Amlodipine/Telmisartan Combined or Alone and Select Better Dose of CKD-828 in Patients With Essential Hypertension
Brief Title: CKD-828 Primary Hypertension Trial(Dose-selection)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Jin Kim / Director
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 128HT09K
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: CKD-828; Hypertension; Primary Hypertension; S-Amlodipine; Telmisartan; Amlodipine; Factorial; Phase 2
MeSH Terms: conditions — Hypertension; Essential Hypertension | interventions — levamlodipine; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (9):
- S-Amlodipine 2.5mg + Telmisartan 40mg (Experimental)
  Interventions: Drug: S-Amlodipine, Telmisartan
- S-Amlodipine 2.5mg + Telmisartan 80mg (Experimental)
  Interventions: Drug: S-Amlodipine, Telmisartan
- S-Amlodipine 5mg + Telmisartan 40mg (Experimental)
  Interventions: Drug: S-Amlodipine, Telmisartan
- S-Amlodipine 5mg + Telmisartan 80mg (Experimental)
  Interventions: Drug: S-Amlodipine, Telmisartan
- S-Amlodipine 2.5mg (Active Comparator)
  Interventions: Drug: S-Amlodipine
- S-Amlodipine 5mg (Active Comparator)
  Interventions: Drug: S-Amlodipine
- Telmisartan 40mg (Active Comparator)
  Interventions: Drug: Telmisartan
- Telmisartan 80mg (Active Comparator)
  Interventions: Drug: Telmisartan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: S-Amlodipine, Telmisartan
  Arms: S-Amlodipine 2.5mg + Telmisartan 40mg; S-Amlodipine 2.5mg + Telmisartan 80mg; S-Amlodipine 5mg + Telmisartan 40mg; S-Amlodipine 5mg + Telmisartan 80mg
Drug: S-Amlodipine
  Arms: S-Amlodipine 2.5mg; S-Amlodipine 5mg
Drug: Telmisartan
  Arms: Telmisartan 40mg; Telmisartan 80mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The aim of this trial is to determine the best dose combination of S-Amlodipine and Telmisartan as compared to monotherapy by assessing the blood pressure lowering effects of a once daily regimen of various combinations of S-Amlodipine and Telmisartan, compared to their monotherapy components and placebo, in patients with stage I or II essential hypertension(a mean seated cuff diastolic blood pressure >=95 and <=115 mmHg).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older
* stage I or II hypertension defined as: a mean seated cuff diastolic blood pressure >=95 and <=115 mmHg
* ability to provide written informed consent

Exclusion Criteria:

* severe hypertension defined as: a mean seated cuff diastolic blood pressure >=116mmHg or a mean seated cuff systolic blood pressure >=200mmHg
* known or suspected secondary hypertension(ex. aortic coarctation, Primary hyperaldosteronism, renal artery stenosis, pheochromocytoma)
* has severe heart disease(Heart failure NYHA functional class 3, 4), unstable angina or myocardial infarction, arrhythmia within the past three months
* has cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months
* Type I Diabets Mellitus, Type II Diabetes Mellitus with poor glucose control as defined by fasting glucosylated hemoglobin(HbA1c) > 8%
* known severe or malignant retinopathy
* hepatic or renal dysfunction as defined by the following laboratory parameters: AST/ALT > UNL X 2, serum creatinine > UNL X 1.5
* acute or chronic inflammatory status need to treatment
* need to additional antihypertensive drugs during the study
* need to concomitant medications known to affect blood pressure during the study
* history of angioedema related to ACE inhibitors or Angiotensin II Receptor Blockers
* known hypersensitivity related to either study drug
* history of drug or alcohol dependency
* any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of investigational products(ex. gastrointestinal tract surgery such as gastrectomy, gastroenterostomy or bypass, active inflammatory bowel syndrome within 12 months prior to screening, currently active gatritis, ulcers of gastrointetinal/rectal bleeding, impaired pancreatic fuction such as pancreatitis,obstructions of the urinary tract or difficulty in voiding)
* cannot swallow investigational products
* administration of other study drugs within 4 weeks prior to randomization
* premenopausal women(last menstration < 1year) not using adequte contraception, pregnant or breast-feeding
* history of malignancy including leukemia and lymphoma within the past 5 years
* in investigator's judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 430 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure(MSDBP) | After 8 weeks of treatment

SECONDARY OUTCOMES:
Mean Sitting Diastolic Blood Pressure(MSDBP) | After 4 weeks of treatment
Mean Sitting Systolic Blood Pressure(MSSBP) | After 4 weeks and 8 weeks of treatment
Response rate | After 4 weeks and 8 weeks of treatment
  Reduction of SBP ≥ 20mmHg, DBP ≥ 10mmHg
Control rate | After 4 weeks and 8 weeks of treatment
  Reduction SBP < 140mmHg, DBP < 90mmHg

CONTACTS AND LOCATIONS:
Locations (26):
- South Korea (26):
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang University Hospital in Bucheon, Bucheon-si
  - Kosin University Gospel Hospital, Busan
  - Chungbuk National Uiversity Hospital, Cheongju-si
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - DonGuk University International Hospital, Goyang
  - National Health Insurance Corporation Ilsan Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Inchon
  - Chonbuk National University Hospital, Jeonju
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Ewha Womans University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kandong Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - Seoul St. Mary's Hospital, The catholic University of Korea, Seoul
  - Severance Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Soon Chun Hyang University Hospital, Seoul
  - St. Paul's Hospital, The catholic University of Korea, Seoul
  - Ajou University Hospital, Suwon
  - Uijeongbu St. Mary's Hospital, The catholic University of Korea, Uijeongbu-si
  - Wonju Christian Hospital, Wŏnju